CLINICAL TRIAL: NCT01505972
Title: Time Schedules for Sending Invitations to Colonoscopy Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NR13002404_1
Record Dates: First submitted 2011-12-08; First posted 2012-01-09 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer
Keywords: screening colonoscopy; attendance; response; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Six and three time schedule (Experimental)
  Interventions: Other: Six and three time schedule
- Four and two time schedule (Experimental)
  Interventions: Other: Four and two time schedule

INTERVENTIONS:
Other: Six and three time schedule — Invitation letter sent 6 weeks and reminder 3 weeks before a pre-specified screening colonoscopy appointment date.
  Arms: Six and three time schedule
Other: Four and two time schedule — Invitation letter and reminder sent 4 and 2 weeks before pre-specified screening colonoscopy appointment date.
  Arms: Four and two time schedule

SUMMARY:
The attendance rate to population based primary screening colonoscopy within NordICC trial (The Nordic-European Initiative on Colorectal Cancer, NCT00883792) in Poland is roughly 33%. The aim of this study is to compare the effect of two different time schedules for sending invitations and reminding letters to a pre-specified colonoscopy appointment. 1,600 screening naive men and women 55 to 64 years of age are randomly assigned in a 1:1 ratio to receive invitation and reminder 6 and 3 weeks (SIX and THREE group) or 4 and 2 weeks (FOUR and TWO group) prior to pre-specified screening colonoscopy appointment date. Outcome measures are participation in screening colonoscopy within 6 months from the date of invitation, response and acceptance rate before sending a reminder. The study is powered to detect 7% difference in participation in screening colonoscopy.

ELIGIBILITY:
Inclusion criteria:

Individuals aged 55-64 years living in Warsaw area randomly drawn from Population Registry and randomized to the screening arm of the NordICC trial.

Exclusion criteria:

* Resident abroad
* Return of unopened letter of invitation and/or reminder (address unknown)
* Message from neighbour/family/post office on death of screenee (not updated in Population Registry).

Exclusion criteria for colonoscopy:

* Individuals with previous colorectal surgery (resections, enterostomies)
* Individuals in need of long-lasting attention and nursing services (somatic or psychosocial, mental retardation).
* On-going cytotoxic treatment or radiotherapy for malignant disease
* Severe chronic (longer than trial duration) cardiac (NYHA III-IV)or lung disease
* Lifelong anticoagulant therapy with Warfarin
* A coronary event requiring hospitalization during the last 3 months
* A cerebrovascular event during the last 3 months

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1600 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Participation rate | 6 months from the date of sending invitation letter
  Percentage of attenders to screening colonoscopy.

SECONDARY OUTCOMES:
Acceptance rate in SIX &THREE group | 3 weeks from the date of sending invitation letter
  Percentage of invitees who agreed (by phone or letter) to participate in screening colonoscopy before sending a reminder
Acceptance rate in FOUR&TWO group | 2 weeks from the date of sending invitation letter, respectively
  Percentage of invitees who agreed (by phone or letter) to participate in screening colonoscopy before sending a reminder
Response rate in SIX&THREE group | 3 weeks from the date of sending invitation letter
  Percentage of invitees who responded (by phone or letter) before sending a reminder
Response rate in FOUR&TWO group | 2 weeks from the date of sending invitation letter
  Percentage of invitees who responded (by phone or letter) before sending a reminder

CONTACTS AND LOCATIONS:
Overall Officials: Regula Jaroslaw, MD, PhD, Study Director — Center of Oncology UInstitute and the Maria Sklodowska-Curie; Kaminski F Michal, MD, Study Chair — Center of Oncology Institute and the Maria Sklodowska-Curie; Pisera Malgorzata, Msc, Principal Investigator — Center of Oncology Institute and the Maria Sklodowska-Curie
Locations (1):
- Center of Oncology Institute and the Maria Sklodowska-Curie, Warsaw, W.K.Roentgena, Poland